CLINICAL TRIAL: NCT05305131
Title: Phase II Randomised Trial of Induction Gemcitabine and Cisplatin Versus Gemcitabine, Cisplatin, Pembrolizumab and Bevacizumab (GPPB) in Nasopharyngeal Cancer
Brief Title: Randomised Trial of Induction Gemcitabine and Cisplatin Versus Gemcitabine, Cisplatin, Pembrolizumab and Bevacizumab (GPPB) in Nasopharyngeal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP01/04/21
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Cancer
Keywords: gemcitabine; cisplatin; pembrolizumab; bevacizumab; GPPB
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Cisplatin; Gemcitabine; Bevacizumab; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This will be a single-centre, open label, randomised phase II study of induction cisplatin and gemcitabine with or without bevacizumab in patients with locally advanced or metastatic NPC. 50 Eligible patients will be randomised 1:1 into either of the two study arms: induction chemotherapy cisplatin and gemcitabine, or induction chemotherapy cisplatin, gemcitabine, bevacizumab and pembrolizumab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Induction cisplatin and gemcitabine (Experimental): Each treatment cycle is 3 weeks. All patients would receive 3 cycles of induction chemotherapy as part of the study, and would then be considered for subsequent concurrent chemoradiotherapy at the investigator's discretion. Cross over is not allowed.
  Interventions: Drug: cisplatin and gemcitabine
- induction chemotherapy cisplatin, gemcitabine, bevacizumab and pembrolizumab (Experimental): Each treatment cycle is 3 weeks. All patients would receive 3 cycles of induction chemotherapy as part of the study, and would then be considered for subsequent concurrent chemoradiotherapy at the investigator's discretion. Cross over is not allowed.
  Interventions: Drug: induction chemotherapy cisplatin, gemcitabine, bevacizumab and pembrolizumab.

INTERVENTIONS:
Drug: cisplatin and gemcitabine — Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2 Day 8: IV Gemcitabine 1000mg/m2
  Arms: Induction cisplatin and gemcitabine
Drug: induction chemotherapy cisplatin, gemcitabine, bevacizumab and pembrolizumab. — Day -7 (+/-1 day): IV bevacizumab 7.5mg/kg diluted in normal saline over 30 minutes Day 1: IV Gemcitabine 1000mg/m2 + IV Cisplatin 75mg/m2+ IV pembrolizumab 200mg over 30 minutes Day 8: IV Gemcitabine 1000mg/m2 Day 15 (for cycles 1 and 2 only): IV bevacizumab 7.5mg/kg diluted in normal saline over 30 minutes
  Arms: induction chemotherapy cisplatin, gemcitabine, bevacizumab and pembrolizumab

SUMMARY:
The investigators hypothesize that the addition of bevacizumab and pembrolizumab to induction cisplatin and gemcitabine is tolerable and improves metabolic complete response (mCR), relapse free survival (RFS) and overall survival (OS) compared to induction cisplatin and gemcitabine in patients with locally advanced nasopharyngeal cancer (NPC)

DETAILED DESCRIPTION:
NPC is endemic in Singapore and southern China, where the southern Chinese have the highest incidence of NPC worldwide.

Nasopharyngeal cancer usually presents as locally advanced stage III or IV disease with T3-4 or N2-3 nodal status.The standard of care of patients with locally advanced NPC is concurrent cisplatin chemotherapy with radiation therapy. However, a significant proportion of patients (about 30% in most randomised phase III studies) still relapse, compromising their survival from NPC. This is particularly so in patients with stage IVA, T4 or N3 NPC. Emerging evidence suggests induction chemotherapy improves patient survival in this group of patients when integrated with concurrent chemoradiation. A meta-analysis also showed that the addition of induction chemotherapy improved overall survival, and reduced locoregional and distant failure.

Dysregulation of the vascular endothelial growth factor (VEGF)/VEGF receptor-2 axis is a feature of many cancers including NPC. Elevated VEGF expression promotes disorganised tumour neovascularisation with hyperpermeable, tortuous capillaries.9, 10 Leakiness of vessels increases interstitial fluid pressure that collapses vessels with the collective effect of compromising blood flow and perfusion, limiting the delivery of therapeutic drugs. Furthermore, tumour expression of VEGF promotes immune tolerance directly and through hypoxic mechanisms.11 The VEGF/VEGFR-2 axis can be inhibited humanised monoclonal antibody bevacizumab, which binds to VEGF-A and prevents ligand-receptor engagement.

As NPC is associated with EBV antigen expression and is characterised by a prominent inflammatory infiltrate (inflammatory immune phenotype), there has been great interest in studying the effect of immune checkpoint inhibitors in NPC. Recently, the addition of 2 antiPD1 monoclonal antibodies, toripalimab 12 and camrelizumab 13, to cisplatin and gemcitabine was studied in 2 phase III trials conducted in mainland China. Both studies demonstrated that addition of antiPD1 therapy to cisplatin/gemcitabine chemotherapy improved the response rate, PFS and the duration of response in treatment naïve patients with metastatic or recurrent NPC.

The investigators have conducted a prior study evaluating pembrolizumab with and without bevacizumab. Preliminary analysis showed a higher response rate for addition of bevacizumab to pembrolizumab compared to pembrolizumab alone arm with no new safety signal. Importantly, the adverse effects of anti-angiogenic and anti PD1 therapy in humans are non-overlapping with cytotoxic chemotherapy. In view of this, investigators are conducting an open label, phase II randomised controlled trial comparing induction cisplatin, gemcitabine, bevacizumab and pembrolizumab with the standard arm (induction cisplatin and gemcitabine) in patients with stage III-IVA locally advanced EBER positive nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The participant (or legally acceptable representative if applicable) provides written consent for the trial.
2. Participants who are at least 21 years of age on the day of signing informed consent with histologically or cytologically confirmed diagnosis of non-keratinizing nasopharyngeal carcinoma (NPC).
3. Have measurable disease based on RECIST 1.1.
4. Tumour stage III (except for T3N0 and T3N1) or IVA according to the American Joint Committee on Cancer (AJCC) 8th edition criteria.
5. Have locally or centrally determined EBV-positive NPC by EBV-encoded small RNA in situ hybridization (EBER in situ hybridization [ISH]) assay. If EBV-positive status has been previously determined by EBER ISH assay, then no re-testing is required.

   Note: If EBV status by EBER ISH assay has not been previously determined, tumor tissue from archival tissue may be submitted for EBV determination.
6. Did not receive any prior treatment
7. Willingness to donate blood for mandatory translational research studies.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Have an adequate organ function
10. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 of study protocol OR
    2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 of study protocol during the treatment period and for at least 120 days after the last dose of study medication.
11. A male participant must agree to use a contraception as detailed in Appendix 3 of study protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

1. Stage III NPC with T3N0 or T3N1 staged by AJCC 8th edition
2. Has received prior systemic anti-cancer therapy including chemotherapy, radiotherapy, immunotherapy or investigational agents
3. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to first dose of study treatment.
4. Has a condition requiring systemic steroid therapy (> 10 mg daily prednisone equivalents) or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if < or = 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
5. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment.
6. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
7. Has hypersensitivity to bevacizumab or any of its components.
8. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

   Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, transitional cell carcinoma of urothelial cancer, or carcinoma in situ (e.g. breast or cervical carcinoma in situ) that have undergone potentially curative therapy are not excluded.
9. Has an active infection requiring systemic therapy, or serious non-healing wound, ulcer or bone fracture.
10. Uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of = 3 anti-hypertensive drugs or systolic blood pressure greater than 150 mmHg).
11. History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) Class II; active coronary artery disease (unstable angina [anginal symptoms at rest] or new-onset angina [began within the last 3 months] or myocardial infarction within the past 6 months). Cardiac arrhythmias requiring anti-arrhythmic therapy (ß-blockers or digoxin are permitted).
12. Persistent proteinuria of NCI-CTCAE Grade 3 or higher (> 3.5 g/24 hours, measured by urine protein/creatinine ratio on a random urine sample).
13. Clinically significant bleeding (NCI-CTCAE Grade 3 or higher) within 30 days prior to start of study medication.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
17. A WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization/allocation (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

    Note: In the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
18. Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
19. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.

    Note: No testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
20. Has received a live vaccine within 30 days of prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine.

Note: Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 21 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
metabolic complete response assessed using FDG PET whole body scan at 12 weeks of assessment using PERCIST 1.0 | up to 3 years

SECONDARY OUTCOMES:
Number of participant with treatment related toxicities | up to 3 years
  Safety of induction cisplatin, gemcitabine, pembrolizumab and bevacizumab, compared to induction cisplatin and gemcitabine, using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Best objective response rate (ORR) as assessed using Response Evaluation Criteria in Solid Tumour (RECIST 1.1) | up to 3 years
Disease free survival (DFS) of patients as defined as the time from initiation of treatment to disease recurrence, or death. | up to 3 years
Overall survival of patients, as defined as the time from initiation of treatment to death. | up to 3 years
Plasma EBV DNA levels and correlation with clinical response to induction treatment | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu MC, Yuan JM. Epidemiology of nasopharyngeal carcinoma. Semin Cancer Biol. 2002 Dec;12(6):421-9. doi: 10.1016/s1044579x02000858. PMID 12450728
- [Background] Petersson F. Nasopharyngeal carcinoma: a review. Semin Diagn Pathol. 2015 Jan;32(1):54-73. doi: 10.1053/j.semdp.2015.02.021. Epub 2015 Feb 25. PMID 25769204
- [Background] Wei WI, Sham JS. Nasopharyngeal carcinoma. Lancet. 2005 Jun 11-17;365(9476):2041-54. doi: 10.1016/S0140-6736(05)66698-6. PMID 15950718
- [Background] Chan KCA, Woo JKS, King A, Zee BCY, Lam WKJ, Chan SL, Chu SWI, Mak C, Tse IOL, Leung SYM, Chan G, Hui EP, Ma BBY, Chiu RWK, Leung SF, van Hasselt AC, Chan ATC, Lo YMD. Analysis of Plasma Epstein-Barr Virus DNA to Screen for Nasopharyngeal Cancer. N Engl J Med. 2017 Aug 10;377(6):513-522. doi: 10.1056/NEJMoa1701717. PMID 28792880
- [Background] Lee AW, Ma BB, Ng WT, Chan AT. Management of Nasopharyngeal Carcinoma: Current Practice and Future Perspective. J Clin Oncol. 2015 Oct 10;33(29):3356-64. doi: 10.1200/JCO.2015.60.9347. Epub 2015 Sep 8. PMID 26351355
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Zhang B, Li MM, Chen WH, Zhao JF, Chen WQ, Dong YH, Gong X, Chen QY, Zhang L, Mo XK, Luo XN, Tian J, Zhang SX. Association of Chemoradiotherapy Regimens and Survival Among Patients With Nasopharyngeal Carcinoma: A Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Oct 2;2(10):e1913619. doi: 10.1001/jamanetworkopen.2019.13619. PMID 31626318
- [Background] Goel S, Duda DG, Xu L, Munn LL, Boucher Y, Fukumura D, Jain RK. Normalization of the vasculature for treatment of cancer and other diseases. Physiol Rev. 2011 Jul;91(3):1071-121. doi: 10.1152/physrev.00038.2010. PMID 21742796
- [Background] Jain RK. Normalization of tumor vasculature: an emerging concept in antiangiogenic therapy. Science. 2005 Jan 7;307(5706):58-62. doi: 10.1126/science.1104819. PMID 15637262
- [Background] Fukumura D, Kloepper J, Amoozgar Z, Duda DG, Jain RK. Enhancing cancer immunotherapy using antiangiogenics: opportunities and challenges. Nat Rev Clin Oncol. 2018 May;15(5):325-340. doi: 10.1038/nrclinonc.2018.29. Epub 2018 Mar 6. PMID 29508855
- [Background] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi YR, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Liu Z, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Feng H, Yao S, Keegan P, Xu RH. Toripalimab or placebo plus chemotherapy as first-line treatment in advanced nasopharyngeal carcinoma: a multicenter randomized phase 3 trial. Nat Med. 2021 Sep;27(9):1536-1543. doi: 10.1038/s41591-021-01444-0. Epub 2021 Aug 2. PMID 34341578
- [Background] Yang Y, Qu S, Li J, Hu C, Xu M, Li W, Zhou T, Shen L, Wu H, Lang J, Hu G, Luo Z, Fu Z, Qu S, Feng W, Chen X, Lin S, Zhang W, Li X, Sun Y, Lin Z, Lin Q, Lei F, Long J, Hong J, Huang X, Zeng L, Wang P, He X, Zhang B, Yang Q, Zhang X, Zou J, Fang W, Zhang L. Camrelizumab versus placebo in combination with gemcitabine and cisplatin as first-line treatment for recurrent or metastatic nasopharyngeal carcinoma (CAPTAIN-1st): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2021 Aug;22(8):1162-1174. doi: 10.1016/S1470-2045(21)00302-8. Epub 2021 Jun 23. PMID 34174189